CLINICAL TRIAL: NCT05990985
Title: A Clinical Study Was Conducted to Evaluate the Efficacy and Safety of the RCMOP Regimen Sequential Therapy as a First-line Treatment for Patients With Intermediate-to-high Risk Diffuse Large B-cell Lymphoma Who Had Incomplete Remission.
Brief Title: The Efficacy and Safety of the RCMOP Sequential Therapy as a First-line Treatment for Patients With Intermediate-to-high Risk Diffuse Large B-cell Lymphoma Who Had Incomplete Remission.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ou Bai, MD/PHD, Director, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-DLBCL-K10
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RCMOP (Experimental): RiTUXimab Injection+Cyclophosphamid+Mitoxantrone hydrochloride liposome injection+Vincristine+Prednisolone, 4 cycles of treatment
  Interventions: Drug: Mitoxantrone hydrochloride liposome injection; Drug: RiTUXimab Injection; Drug: Cyclophosphamid; Drug: Vincristine; Drug: Prednisolone

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome injection — Mitoxantrone hydrochloride liposome injection (18 mg/m^2) will be administered by intravenous infusion on day 1 in a 3-week treatment cycle.
  Other Names: duoenda
Drug: RiTUXimab Injection — RiTUXimab Injection (375 mg/m^2) will be administered by intravenous infusion on day 0 in a 3-week treatment cycle.
  Other Names: lituoxidankang
Drug: Cyclophosphamid — Cyclophosphamid (750 mg/m^2) will be administered by intravenous infusion on day 1 in a 3-week treatment cycle.
  Other Names: huanlinxianan
Drug: Vincristine — Vincristine (1.4 mg/m^2，maximum dose 2mg ) will be administered by intravenous infusion on day 1 in a 3-week treatment cycle.
  Other Names: changchunxinjian
Drug: Prednisolone — Prednisolone (100mg/d) will be administered by intravenous infusion on day 1-5 in a 3-week treatment cycle.
  Other Names: ponisong

SUMMARY:
A clinical study was conducted to evaluate the efficacy and safety of the RCMOP regimen sequential therapy as a first-line treatment for patients with intermediate-to-high risk diffuse large B-cell lymphoma who had incomplete remission.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent
2. Age≥18 years old
3. International Prognostic Index (IPI)>2
4. Expected survival ≥ 3 months
5. DLBCL initially diagnosed by histopathology meets the following subtypes according to the 2016 WHO classification: (1) Germinal center B-cell-like (GCB) subtype; (2) Non-germinal center B-cell-like (non-GCB) subtype
6. Patients who were evaluated as incomplete remission after 2 cycles of RCHOP/RCDOP for initial treatment
7. At least 1 evaluable or measurable lesion meeting Lugano 2014 criteria: Nodal lesion: Greatest transverse diameter>1.5cm; Extra-nodal lesion: Greatest transverse diameter>1.0cm
8. ECOG Performance Status: 0-1
9. Bone marrow function: Absolute neutrophil count ≥1.5×10^9/L, Platelet count ≥75×10^9/L, Hemoglobin ≥ 80g/L (Patients with bone marrow involvement were judged by the investigator to enter the group)
10. Liver and kidney function: serum creatinine ≤ 1.5×ULN (upper limit of normal); AST and ALT ≤ 2.5×ULN (≤ 5×ULN for subjects with liver metastases); total bilirubin ≤ 1.5×ULN (≤ 3×ULN for subjects with liver metastases).

Exclusion Criteria:

1. Hypersensitivity to any study drug or its components
2. Uncontrolled systemic diseases (such as active infection, uncontrolled hypertension, diabetes, etc.)
3. Heart function and disease meet one of the following conditions: (1) Long QTc syndrome or QTc interval > 480 ms; (2) Serious and uncontrolled arrhythmias requiring drug treatment, uncontrolled angina with poor drug control and myocardial infarction within 6 months before enrollment; (3) New York Heart Association grade III~IV; (4) Cardiac ejection fraction (LVEF)< 45%
4. Hepatitis B and hepatitis C active infection (HBV DNA above upper limit of normal; HCV antibody positive and HCV RNA above upper limit of normal)
5. Human immunodeficiency virus (HIV) infection (HIV antibody positive)
6. Subjects with other malignant tumors past or present (except for non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in control, and other malignant tumors that have been effectively controlled without treatment within the past five years)
7. Subjects suffering from primary or secondary central nervous system (CNS) lymphoma
8. pregnancy, lactation and patients of childbearing age who are unwilling to take contraceptive measures
9. Mental patients or those who cannot obtain informed consent
10. Unsuitable subjects for this study determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of cycle 2, At the end of cycle 4, (each cycle is 21 days)
  To evaluate the efficacy of anti-tumor

SECONDARY OUTCOMES:
Complete response rate (CRR) | At the end of cycle 2, At the end of cycle 4; (each cycle is 21 days)
  To evaluate the efficacy of anti-tumor
Duration of Response (DOR) | CR or PR up to data cut-off (up to approximately 2 years)
  To evaluate the efficacy of anti-tumor
Progression-free survival (PFS) | Baseline up to data cut-off (up to approximately 2 years)
  To evaluate the efficacy of anti-tumor
Overall survival (OS) | Baseline up to data cut-off (up to approximately 2 years)
  To evaluate the efficacy of anti-tumor
Treatment emergent adverse events (TEAEs) | The first dose up to 21 or 28 days after the last dose
  The incidence and severity of adverse events assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China